CLINICAL TRIAL: NCT04861844
Title: Tracking Mood and Language Change Across a Phone-based Mindfulness Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty recruiting patients, staffing
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sara Bradley, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00214284
Record Dates: First submitted 2021-03-08; First posted 2021-04-27 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness training (Experimental)
  Interventions: Behavioral: mindfulness training
- Active listening (Active Comparator)
  Interventions: Behavioral: active listening

INTERVENTIONS:
Behavioral: mindfulness training — phone based mindfulness training on 4 consecutive days
  Arms: Mindfulness training
Behavioral: active listening — The active listening intervention script asks the participant to attend by relaxing their body and visualizing themself in various exotic locations and narratives described in the script; it also asks the participant to rate their attention level of various points. The active listening scripts were compiled from National Geographic article excerpts (taken from the public domain)
  Arms: Active listening

SUMMARY:
The objective of this study is to administer a brief, phone(voice)-based training program in mindfulness (or control task of active listening to narrated articles) to older adults who receive primary care services at NM. Older adults represent a population that is at risk for depression and anxiety, especially during the current COVID-19 pandemic and the social isolation it entails. Many older adults also possess relatively low access to application-based mindfulness training opportunities. The monitoring aims are:

1. To determine whether the experimental intervention (mindfulness training) performs better than a control task (active listening) in improving mood assessed using the Profile of Mood States (POMS) and/or anxiety assessed using the State-Trait Anxiety Inventory (STAI).
2. To determine whether the experimental and/or control intervention is associated with quantified changes in language use (e.g., frequency of negative word use), which may or may not also be associated with changes in mood and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients part of the Northwestern Medicine Geriatrics Practice, or Northwestern Feinberg School of Medicine ECMH program.
2. English-speaking; and
3. Able to verbally consent

Exclusion Criteria:

patients with dementia or otherwise not meeting inclusion criteria

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Change in mood assessed using the Profile of Mood States (POMS) | 3 days
  The Profile of Mood States (POMS) is a widely used instrument that measures mood using a 65-item questionnaire with each item rated using a response scale of five categories ranging from "not at all" to "very strong". Higher score indicates worse mood.
Change in anxiety assessed using the State-Trait Anxiety Inventory (STAI). | 3 days
  The State-Trait Anxiety Inventory (STAI) is psychological inventory consisting of 40 questions rated on a 4-point Likert scale. Higher score correlates with higher levels of anxiety.
Change in mood assessed using the Profile of Mood States (POMS) | 1 month
  The Profile of Mood States (POMS) is a widely used instrument that measures mood using a 65-item questionnaire with each item rated using a response scale of five categories ranging from "not at all" to "very strong". Higher score indicates worse mood.
Change in anxiety assessed using the State-Trait Anxiety Inventory (STAI). | 1 month
  The State-Trait Anxiety Inventory (STAI) is psychological inventory consisting of 40 questions rated on a 4-point Likert scale. Higher score correlates with higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided